CLINICAL TRIAL: NCT05880472
Title: Percutaneous Intratumoural Holmium Microspheres Brachytherapy for Patients With Pancreatic Cancer; a Single Centre, Prospective Safety and Feasibility Study
Brief Title: Percutaneous Holmium Injection in Pancreatic Cancer
Acronym: SLOTH-2a
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Quirem Medical B.V. (Industry); Terumo Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL.82292.091.22
Record Dates: First submitted 2023-05-09; First posted 2023-05-30 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Pancreas Cancer
Keywords: Intratumoral therapy; Brachytherapy; Holmium-166; Holmium-166 microspheres
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental): Single or multiple injections of holmium-166 microspheres (up to 150 Gy) in a single session. Intervention is not repeated.
  Interventions: Device: Intratumoral

INTERVENTIONS:
Device: Intratumoral — Comparable to CE-marked QuiremSpheres(R) outside of intended use with minor altered specification.
  Other Names: Intratumoural holmium-166 microspheres

SUMMARY:
This investigator initiated study with a medical device aims to assess the safety and feasibility of percutaneous injected holmium-166 microsphere brachytherapy in patients with irresectable pancreatic cancer.

DETAILED DESCRIPTION:
Objective: To test the feasibility and safety of minimally invasive CT-guided percutaneous holmium-166 microsphere brachytherapy in patients suffering from irresectable pancreatic cancer. Study design: This is a single centre, prospective, safety and feasibility study with a medical device in a maximum of 6 patients.

Study population: Patients diagnosed with pathologically proven pancreatic adenocarcinoma, who are ineligible for exploratory surgery or surgical resection of the tumour after 8 cycles of systemic therapy or less in case of unacceptable toxicity, patient refusal or patients who are ineligible for systematic therapy.

Intervention (if applicable): A radioactive medical device will be implanted by CT-guided percutaneous injection. The medical device in question are beta-minus (β-) and gamma(γ) emitting holmium-166 poly(L-lactic acid) microspheres (166Ho-PLLA-MS, HoMS) in a 0.1% Pluronic or cellulose based suspension.

Main study parameters/endpoints: The main endpoint is to establish the feasibility and safety of CT-guided percutaneous intratumoural implantation of HoMS in irresectable pancreatic adenocarcinoma. Feasibility is established by evaluating the average tumour absorbed dose in Gray (Gy) calculated on SPECT and comparing to the pre-operative planning. Intratumoural microsphere distribution, absorbed tumour dose and non-target absorbed tumour dose are analysed using MRI and CT quantification. Safety is evaluated using the Common Terminology Criteria for Adverse Events (CTCAE v5.0), events deemed 'unlikely', 'probably' or 'definitely' related to the implantation procedure or implanted medical device. As exploratory endpoints, tumour response (RECIST1.1), pain (NRS) and Quality of Life is evaluated. Total follow-up is 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged 18 years and over.
2. Pathologically proven pancreatic adenocarcinoma, also known as pancreatic ductal adenocarcinoma.
3. Patient is deemed ineligible for surgical resection of the pancreatic cancer:

   1. in accordance with consensus at the multidisciplinary meetings/discussions,
   2. and/or the patient refuses to undergo surgical resection out of personal choice
4. Life expectancy of 16 weeks or longer.
5. World Health Organisation (WHO) Performance status 0-1
6. One or more measurable pancreatic tumours of at least 20 mm in the longest diameter by spiral CT or MRI according to the Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria.
7. Negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

1. Radiation therapy within the last 4 weeks before the start of study therapy.
2. Chemotherapy within the last 2 weeks before the start of study therapy.
3. Calcifications in the pancreas or tumour that are highly expected to obstruct the needle tract
4. Any unresolved toxicity ≥ grade 3 from the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE version 5.0) from previous anti-cancer therapy.
5. Leukocytes < 3.0 10^9/l and/or platelet count < 75 10^9/l.
6. Kidney failure: Creatine > 165 µmol/l and/or eGFR < 60 ml/min/1,73m^2
7. Significant cardiac event (e.g. myocardial infarction, superior vena cava (SVC) syndrome, New York Heart Association (NYHA) classification of heart disease ≥2 within 3 months before entry, or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
8. Patient is deemed ineligible for implantation of 166Ho by an expert panel (surgeon, nuclear medicine physician, interventional radiologist, radiologist, and researcher) due to tumour anatomy, nearby structures, patient status or a combination.
9. Pregnancy or breast feeding (women of child-bearing potential).
10. Patients suffering from psychic disorders that make a comprehensive judgement impossible, such as psychosis, hallucinations and/or depression.
11. Patients who are declared incompetent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-04-22 (Estimated); Study Completion 2025-04-22 (Estimated)

PRIMARY OUTCOMES:
Average tumour dose (Gy) by SPECT/CT | Within 24 hours post-intervention
  Tumour and non-tumour dose is estimated by SPECT using after intervention to assess feasibility.
Number of adverse event per patient per grade by CTCAE v5.0 | Up to 16 weeks post-intervention
  Number and grade of adverse events per patient by Common Terminology Criteria for Adverse Events (CTCAE v5.0) between grade 0 (mild complication) to grade 5 (death) deemed 'unlikely', 'probably', or 'definitely' related to the implantation procedure or medical device implanted.

SECONDARY OUTCOMES:
Average tumour dose (Gy) by MRI quantification | <24 hour and 16 weeks post-intervention
Average tumour dose (Gy)by CT quantification | <24 hour and 16 weeks post-intervention
Microsphere distribution (percentage covered) of 3D target area | <24 hour and 16 weeks post-intervention
  By CT or MRI to assess dose coverage
Injection percentage (%) | Immediately after the intervention
  Implant efficiency
Needle tip position off-target (mm) | Immediately after the intervention
  implant accuracy
Operator hand and total body dose (mSv) | Immediately after the intervention
  Operator safety

OTHER OUTCOMES:
Tumor response by RECIST 1.1 | 16 weeks post-intervention
  Tumor response by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST). Response is categorised by complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD).
Pain-scale assessment by Numeric Pain Rating Scale (NRS) | Up to 16 weeks post-intervention
  Numeric (Pain) Rating Scale from average and worst pain in past week with 0 = no pain and 10 = worst possible pain
Implantation experience by questionnaire to the operator | Immediately after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Frank Nijsen, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided